CLINICAL TRIAL: NCT02764177
Title: Effect of Recovery Drink Composition Consumed After Resistance Exercise on Subsequent Appetite and Energy Intake
Brief Title: Resistance Exercise, Recovery Drinks and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Lewis James, Dr Lewis James, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: R15-P106
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Active Population

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein (Experimental): In this arm the subjects were provided with a PROTEIN drink to consume after exercise. This protein drink contained whey protein isolate that provided 0.3 g/ kg body mass of protein.
  Interventions: Dietary Supplement: Protein drink
- Carbohydrate (Experimental): In this arm the subjects were provided with a CARBOHYDRATE drink to consume after exercise. This carbohydrate drink was energy matched to the protein drink in the other arm of the experiment.
  Interventions: Dietary Supplement: Carbohydrate drink

INTERVENTIONS:
Dietary Supplement: Protein drink — The protein drink was administered during this trial
  Arms: Protein
Dietary Supplement: Carbohydrate drink — The carbohydrate drink was administered in this trial
  Arms: Carbohydrate

SUMMARY:
Whilst the effects of manipulating the macronutrient content of foods on appetite and energy intake has been relatively well studied at rest, little is known about these responses in a post-exercise context. The effect of post-exercise nutrition on recovery from or adaptation to exercise has been well studied. However, many exercisers do so for weight management and thus any post-exercise nutrition might impact on energy balance and might need to be carefully considered. This study will examine the impact of manipulating the composition of a recovery drink consumed after resistance exercise on subsequent appetite and energy intake.

DETAILED DESCRIPTION:
Subjects perform a bout of lower body resistance exercise lasting ~50 min and immediately post-exercise they consume one of two recovery drinks over a 5 min period. Over the next 60 min subjective appetite responses will be measured and then 60 min after drink ingestion, subjects will consume an ad-libitum meal.

ELIGIBILITY:
Inclusion Criteria:

* Generally fit and healthy
* Use resistance exercise as part of weekly training
* Weight stable in previous 6 months

Exclusion Criteria:

* Smoker
* History of gastric, digestive, cardiovascular or renal disease
* Lactose, dairy, gluten intolerances or allergies

Ages: 18 Years to 60 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Ad-libitum energy intake | 65 min post-exercise
  Assessed via a homogenous pasta meal
Subjective appetite (hunger) | 150 min
  Assessed via 100 mm visual analogue scales
Subjective appetite (fullness) | 150 min
  Assessed via 100 mm visual analogue scales
Subjective appetite (desire to eat) | 150 min
  Assessed via 100 mm visual analogue scales
Subjective appetite (prospective food consumption) | 150 min
  Assessed via 100 mm visual analogue scales

SECONDARY OUTCOMES:
Pleasantness of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Aftertaste of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Saltiness of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Bitterness of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Sweetness of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Creaminess of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Thickness of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Stickiness of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Fruitiness of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Refreshment of study drinks | Immediately after drinking
  Assessed via 100 mm visual analogue scales
Eating rate | 65 min post-exercise
  mean eating rate determined at ad-libitum meal